CLINICAL TRIAL: NCT07223268
Title: Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation (CARE-D-Foot-Nav)
Brief Title: Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marcos C. Schechter, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008140; 1R01DK139326-01A1 (NIH)
Record Dates: First submitted 2025-10-23; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation; Wound care; Wound healing
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Following discharge, the team will conduct research retention phone calls at 4, 8, 12, 16, and 20 weeks to review resource utilization over the past month.
  Participants will have access to hospital and community resources available to all patients treated within the healthcare system.
  Other resources may include, but are not limited to, social worker assistance with transportation, diabetes education (with referral by medical provider), nutritional support through Grady's "Food as Medicine Program", and interpreter services
  Interventions: Other: Standard of care
- CARE-D-Foot-Nav (Experimental): Participants in this arm will be assigned a dedicated DFU patient navigator The navigators will conduct 30-to 60-minute encounters, either by phone or in person, at least once a week during the 20-week program.
  Participants can call the navigator with DFU-related concerns during the navigator's working hours.
  Interventions: Other: CARE-D-Foot-Nav

INTERVENTIONS:
Other: CARE-D-Foot-Nav — CARE-D-Foot-Nav is a diabetes educator who will serve as a dedicated Diabetic Foot Ulcer (DFU) patient navigator.
  The navigator will assist the subjects with diabetic foot ulcer care, including: Glycemic control, Wound management, Infection management, and peripheral artery disease (PAD) management.
  Apart from that, the navigator will also provide tools to improve access to DFU care and emotional support, like: Outpatient care coordination, Transportation assistance, Language-concordant care, Peer support, Support if amputations are recommended, and Spiritual Support.
  Navigator will also assess the participants and screen for Depression, tobacco use, food insecurity, alcohol use, financial resource strain, and housing instability.
  Arms: CARE-D-Foot-Nav
Other: Standard of care — Standard of care for DFU.
  Arms: Standard of Care

SUMMARY:
The purpose of this interventional study is to assess the effectiveness of CARE-D-Foot, a patient navigator intervention, as compared to usual care, on 20-week diabetic foot ulcer healing.

The study will further:

* Evaluate fidelity to and acceptability of the CARE-D-Foot-Nav program using mixed methods
* Perform a CARE-D-Foot-Nav cost-effectiveness analysis (CEA)

DETAILED DESCRIPTION:
The CARE-D-Foot-Nav (Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation) study is a randomized controlled trial testing whether a patient navigator-led intervention can improve healing outcomes for patients hospitalized with diabetic foot ulcers (DFUs). DFUs are a serious complication of diabetes that contribute to over 100,000 amputations annually in the U.S. and account for a significant portion of diabetes-related healthcare costs. Healing requires complex, multidisciplinary care focused on glycemic control, wound management, vascular disease treatment, and infection therapy. However, many patients, especially underserved populations such as non-Hispanic Black and Hispanic individuals, face barriers related to social determinants of health that hinder access to this care.

In this trial, 270 patients hospitalized with DFUs will be randomized to receive either usual care or participate in the CARE-D-Foot-Nav program for 20 weeks after hospital discharge. Participants in the intervention group will receive weekly support from a certified diabetes educator acting as a patient navigator, who will provide personalized care coordination, diabetes education, transportation assistance, and help connecting patients to medical and social resources.

Navigators have proven effective in improving outcomes for other chronic diseases by overcoming healthcare system and patient-level barriers, but no prior randomized trials have tested their impact on DFU care specifically. This study aims to fill that gap by evaluating whether the CARE-D-Foot-Nav program improves DFU healing rates, enhances patient engagement, and can be implemented cost-effectively. The intervention is designed to be scalable and focused on reducing healthcare disparities to help curb the diabetes-related amputation epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diabetes admitted for any reason who have a full-thickness DFU (defined as a wound below the ankle through the dermis) or undergo a single toe amputation
* History of prior amputations and DFUs of any severity

Exclusion Criteria:

* Adults unable to understand the nature and scope of the study, enrolled in another clinical trial, or planned for discharge to an acute or long-term care facility,
* Patients who undergo amputation of two or more toes during hospitalization and/or have a Society for Vascular Surgery Wound, Ischemia, foot Infection grade 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of CARE-D-Foot-Nav: 20-week wound healing with complete re-epithelialization of the wound | Baseline, Week 20 (day 140 +/- 7 days)
  Pictures will be taken at baseline and week 20 and compared by two different reviewers. The number of participants with complete wound healing will be reported.

SECONDARY OUTCOMES:
Number of participants with confirmed wound healing | Baseline, week 22
  Researchers will measure the effectiveness of the intervention based on wound healing. Photographs of the wounds will be taken at enrollment and again at week 22 (i.e., approximately two weeks ±7 days after the participant's primary outcome visit). Two independent reviewers, who are clinical DFU experts, will evaluate the photographs to determine whether wound healing has occurred.
  If more than one DFU is present, the assessment will be based on the largest wound. If a participant undergoes an amputation or dies before week 20, the ulcer will be classified as not healed.
DFU care clinic attendance | Within 14 and 30 days post hospital discharge
  This will be defined as attending outpatient visits with any provider managing a) diabetes b) wound care c) antibiotic for DFU infection, if applicable, and (d) obtaining non-invasive PAD testing if not done in the last 12 months.
Wound area reduction | Baseline, Week 20
  Difference in diabetic foot ulcer area will be reported
Major amputation | Baseline, Week 20
  Number of subjects undergoing amputation above the ankle.
Number of deaths | Baseline, Week 20
  Number of deaths during the study period.
EuroQol five-dimensional (EQ-5D) score | Baseline, Week 20
  The EuroQol 5-Dimension (EQ-5D) is a standardized instrument used to measure health-related quality of life. It's a self-report questionnaire that assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a few levels of severity, allowing individuals to describe their health state. Each dimension has five levels: 1 = no problems, to 5 = extreme problems/unable to do. The five answers produce a unique 5-digit health state, for example, 11234, that describes the young person's health state. For example, the code 11234 describes a health state where there are no problems with walking about (mobility) or looking after myself, a little bit of a problem with doing usual activities, some pain or discomfort, and feeling really worried, sad, or unhappy.
Glycemic control: Change in HbA1c | Baseline, Week 20
  Change in hemoglobin A1c will be reported.
Perceived social support: Interpersonal Support Evaluation List-12 | Baseline, Week 20
  The Interpersonal Support Evaluation List-12 (ISEL-12) is a brief, validated questionnaire designed to assess perceived availability of social support. The ISEL-12 includes 12 items and evaluates perceived support across three dimensions: Appraisal Support, Belonging Support and Tangible Support.
  Each item is rated on a 4-point Likert scale. Scores range from 12 to 48, with higher scores indicating greater perceived social support and low scores indicating lower social support.
Medical mistrust: Change in the Trust in Physicians Scale | Baseline, Week 20
  Trust in Physicians Scale is used to measure interpersonal trust a patient has in their individual physician.
  Each item is rated on a 5-point Likert scale. Total score range: 11 (low trust) to 55 (high trust).
  Higher scores indicate greater trust in the physician.
Tobacco cessation | Baseline, Week 20
  Self-reported cessation at week 20 among those reporting tobacco use at baseline
Acute care utilization | After hospital discharge (up to 20 weeks)
  All-cause emergency department (ED) visits and re-hospitalizations
Services accessed | Baseline, Week 20
  Services accessed between baseline and week 20 (e.g., foodbank) ascertained through electronic medical record review and participant interviews
Peer support group attendance | Baseline, Week 20
  Proportion of CARE-D-Foot-Nav participants who attended ≥1 peer support group meeting and the number of meetings attended
Diabetic foot ulcer - short form (DFS-SF) score | Baseline, 20 weeks
  A short form of the Diabetic Foot Ulcer Scale (DFS), which is called the Diabetic Foot Ulcer Scale-Short Form (DFS-SF). It's a 29-item questionnaire designed to assess the impact of diabetic foot ulcers on a patient's quality of life (QOL), grouped into six subscales: leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, and bothered by ulcer care. Each item is scored on a 5-point Likert scale, ranging from 1 = "not at all" to 5 = "very common". Each subscale is scored on a scale of 0 to 100. Higher scores on the DFS-SF indicate a better quality of life, while lower scores indicate a poorer quality of life.
  The minimum score for each subscale is 0, representing the worst QOL, and the maximum score is 100, representing the best QOL.
Patient Health Questionnaire-2 (PHQ-2) | Baseline, 20 weeks
  The PHQ-2 is a two-question screening for depression that asks about the frequency of a depressed mood and lack of pleasure in activities over the past two weeks. Scores range from 0 to 6, with a score of 3 or higher indicating a positive screen that warrants further assessment, typically with the full PHQ-9, to confirm a diagnosis and gauge severity.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 20 weeks
  The PHQ-9 is a screening tool for depression that uses nine questions answered on a 0-3 scale (not at all, several days, more than half the days, nearly every day), with the total score ranging from 0 to 27. A professional assesses the total score to gauge depression severity: 0-4 (minimal), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), and 20+ (severe).
Food insecurity | Baseline, Week 20
  Food insecurity will be assessed via validated EHR-embedded survey items. Food insecurity severity is often evaluated based on the number of affirmative responses to specific questions. More affirmative responses typically indicate greater food insecurity.
Housing stability | Baseline, Week 20
  Housing Stability will be assessed using survey items embedded in the electronic health record (EHR). Responses are coded as:
  0 = Stable housing (e.g., own/rent a steady place to live)
  1 = Unstable housing (e.g., temporarily staying with others, in a shelter, or without a place to live) Scores will be summarized as the proportion of participants with unstable housing at baseline and week 20.
Financial resource strain questionnaire | Baseline, Week 20
  Financial resource strain scoring assesses the level of difficulty individuals experience in meeting their basic living expenses and financial obligations, assessed via validated EHR-embedded survey items. A score of 27 on the Financial Strain Questionnaire indicates greater financial strain than a score of 9. Lower scores/categories indicate less financial strain. Higher scores indicate greater strain.
Transportation needs | Baseline, Week 20
  Transportation needs will be assessed via a validated EHR-embedded transportation survey from the Protocol for Responding to and Assessing Patients' Assets, Risks, and Experiences (PRAPARE) tool.
  The transportation tool is a 2-question survey where "yes" indicates transportation needs. More affirmative responses typically indicate increased transportation needs.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Schechter, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The team will de-identify identifiable data and assign each study participant a unique identifier (ID). The team will use the Safe Harbor method to comply with the HIPAA Privacy Rule. The Safe Harbor method removes all 18 identifiers of Protected Health Information (PHI) from data to ensure that the data cannot be traced back to one person. PI will share the individual-participant level raw data described below through deposition in a controlled-access public repository (Emory Dataverse). To preserve participant anonymity and safety, PI will not share participant interviews or navigator encounter audio recordings. We will redact interview transcripts and encounters to remove any potential identifiers. Foot images will be edited to remove identifying features, including faces. The informed consent forms will reflect these plans.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start: January 1, 2031. End: life of the Emory Dataverse Repository
Access Criteria: Requests via email

REFERENCES:
- [Derived] Schechter MC, Rhodes EC, Shao H, Ahmed S, Colquitt K, Chaudhry NY, Dunlop AL, Flores J, Garcia-Toca M, Javia V, Kalokhe AS, Manoj A, Meadows C, Meriwether N, Sales JM, Soleimanmanesh N, Santamarina G, Smith-Bankhead NK, Umpierrez G, Ramos CR, Watson E, Peng L, Fayfman M. A randomized controlled trial of patient navigators for post-hospital discharge diabetic foot ulcer care: the Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation (CARE-D-Foot-Nav) study protocol. medRxiv [Preprint]. 2025 Nov 27:2025.11.25.25340976. doi: 10.1101/2025.11.25.25340976. PMID 41358308